CLINICAL TRIAL: NCT03901924
Title: A Phase III Randomized Trial Comparing the Effects of Volume Support and Assist Control Mode Ventilation on Ventilator-Free Days and Diaphragmatic Atrophy
Brief Title: Volume Support/Assist Control Mode Ventilation and Diaphragmatic Atrophy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-1482
Record Dates: First submitted 2019-02-27; First posted 2019-04-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Mechanical Ventilation Complication
Keywords: Diaphragm Atrophy; Ventilator Induced Diaphragm Dysfunction; Mechanical Ventilation; Volume Support Mode; Assist Control Mode; Diaphragm Thickening Fraction; Intubation; Delirium; Ventilator-Free Days
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor will be masked to randomization and ventilator settings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volume Support Mode Mechanical Ventilation (Active Comparator): Volume support mode ventilation is a spontaneous mode where a target goal volume is set on the ventilator. This ventilatory strategy is dependent on patients spontaneously breathing and triggering (or activating) the ventilator to support the breath. The ventilator adjusts the amount of pressure support to deliver with each breath (i.e. if the patient's tidal volume is greater than the set target volume, then the ventilator will decrease the amount of pressure support in the subsequent breath to try to achieve the goal volume and vice versa). The respiratory rate is not set in this mode of ventilation and is dependent on the patient. For patients randomized to this mode, the goal tidal volume will be set at 6 cc/kg of ideal body weight (IBW).
  Interventions: Other: Volume Support Mode Mechanical Ventilation
- Assist Control Mode Mechanical Ventilation (Active Comparator): In assist control mode ventilation, the machine is programmed to deliver a set tidal volume and set respiratory rate. Patients can breathe over the set respiratory rate, but the volume of breath that they receive is fixed and delivered by the ventilator. For patients randomized to this mode, the tidal volume will be set at 6 cc/kg of ideal body weight (IBW).
  Interventions: Other: Assist Control Mode Mechanical Ventilation

INTERVENTIONS:
Other: Volume Support Mode Mechanical Ventilation — This is a spontaneous mode of mechanical ventilation that depends on the patient's efforts. A target volume (6 cc/kg of IBW), PEEP and FiO2 are set by the medical team, and the ventilator varies the inspiratory pressure support with each breath to achieve the target volume. The respiratory rate is fully dependent on the patient. Sedation while on mechanical ventilation will be set at a goal RASS of 0 to -2.
  Arms: Volume Support Mode Mechanical Ventilation
Other: Assist Control Mode Mechanical Ventilation — This is a controlled mode of mechanical ventilation that is independent of patient's efforts. A tidal volume (6 cc/kg of IBW), respiratory rate, PEEP and FiO2 are set by the medical team. Sedation while on mechanical ventilation will be set at a goal RASS of 0 to -2.
  Arms: Assist Control Mode Mechanical Ventilation

SUMMARY:
The objective of the study is to determine how controlled mode ventilation and support mode ventilation impact ventilator-free days and diaphragmatic atrophy.

DETAILED DESCRIPTION:
Ventilator-induced diaphragmatic dysfunction (VIDD) is characterized by diaphragmatic atrophy and weakness leading to an inability to liberate from the ventilator. Patients with VIDD have increased intensive care unit and hospital length of stay, higher reintubation rates, and need for tracheostomy. There are two commonly used modes of ventilation in the ICU - controlled and support mode ventilation. Conventional practice is to initiate mechanical ventilation with controlled mode followed by a support mode to facilitate weaning and eventual extubation. However, this approach may induce irreversible diaphragmatic atrophy. Observational studies suggest that controlled ventilation is associated with higher rates of diaphragmatic atrophy than support modes of ventilation. Diaphragmatic atrophy occurs within the first 24 hours of mechanical ventilation. To date, it remains unknown whether early initiation of support mode ventilation prevents VIDD and its associated complications in comparison to controlled mode ventilation.

The investigators hypothesize that by initiating subjects on support mode ventilation, an associated increase in ventilator-free days will be seen in comparison to subjects on controlled mode ventilation. Subjects on support mode ventilation will have less diaphragmatic atrophy and weakness than subjects on controlled mode ventilation. To investigate this hypothesis,investigators are conducting a phase III randomized trial examining the effects of volume support mode versus assist control mode ventilation on ventilator-free days and rate of diaphragm atrophy.

enrolled subjects requiring mechanical ventilation will be randomized to either volume support mode or assist control mode within 24 hours of mechanical ventilation initiation. Diaphragm thickness will be measured by ultrasound daily and subsequently diaphragm atrophy rate will be calculated in each arm. The operator acquiring ultrasound images will be blinded to the ventilator mode that the subject was randomized to. Subjects in the study will follow standard ICU sedation awakening trials and spontaneous breathing trials. The medical team in charge of the subject will determine when the subject will be liberated from the ventilator.

There will be up to a 24 hour period from initiation of standard, non-study mechanical ventilation during which the subject can be consented and enrolled. This will allow the research team time to contact the subject and/or family in order to obtain informed consent. Once randomized, all subjects will be initiated on study mode of ventilation. The medical team will direct other aspects of care.

The phase III trial will be powered to determine if there is a statistically significant difference in rate of diaphragm atrophy and ventilator-free days between volume support mode and assist control mode.

ELIGIBILITY:
Inclusion Criteria:

subjects > 18 years of age that have been intubated and mechanically ventilated for < 36 hours at the time of screening will be eligible for enrollment

Exclusion Criteria:

1. pregnancy
2. cardiopulmonary arrest
3. history of diaphragmatic paralysis or neuromuscular disease
4. chronic obstructive pulmonary disease (COPD) or asthma exacerbation with evidence of auto-PEEPing requiring intubation
5. neuromuscular blockade
6. expectation to be liberated from ventilator in < 24 hours
7. history of mechanical ventilation in the last 6 months
8. presence of tracheostomy
9. high cervical spine injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Ventilator-Free Days | 28 days
  A Phase III Primary Outcome; Defined as days alive and free from mechanical ventilation at day 28

SECONDARY OUTCOMES:
Rate of Diaphragm Atrophy | Through study completion, an average of 28 days
  Defined as percentage decline in diaphragm thickness per day

OTHER OUTCOMES:
Noninvasive Measurements of Diaphragm Inspiratory Strength 3.+ 9+ Noninvasive Measurements of Diaphragm Function | Through study completion, an average of 28 days
  negative inspiratory force (nif)--measured unit cm H2O
Noninvasive Measurements of Diaphragm Expiratory Strength | Through study completion, an average of 28 days
  positive expiratory force (pef)--measured unit cm H2O
Diaphragm Thickening Fraction | Through study completion, an average of 28 days
  (diaphragm thickness at end expiration - diaphragm thickness at end inspiration)/diaphragm thickness at end expiration; measured by ultrasound
Duration of Mechanical Ventilation | 28 days
  Days on mechanical ventilation
Frequency of Ventilator-Related Complications | Through study completion, an average of 28 days
  Including the Following: -reintubation
  * tracheostomy
  * mechanical ventilation > 14 days
  * patients with delirium
Readmission to ICU During Same Hospital Admission | Through study completion, an average of 28 days
  Bivariate outcome regarding readmission to ICU--"Yes or No"
Death in ICU | 90 days
  Death that occurs while in the ICU
Death in Hospital | 90 days
  Death that occurs while in the Hospital
Discharge Destination | 90 days
  i.e. home, long term assisted care, skilled nursing facility, death
Mortality | 1 month, 3 months, and 12 months
  measured at 28 days, 90 days, and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Study Director — University of Chicago; Bhakti Patel, MD, Principal Investigator — University of Chicago; Roger Struble, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa